CLINICAL TRIAL: NCT05354024
Title: Phase II/III Double-blind, Randomized Clinical Trial With Active Vaccine Control to Evaluate the Safety, Immunogenicity, and Consistency of the Lots of Booster Dose of COVID-19 (Recombinant, Inactivated) Vaccine in Adults in Brazil
Brief Title: Phase II/III Randomized Clinical Trial of Booster Dose of COVID-19 (Recombinant, Inactivated) Vaccine
Acronym: Butanvac
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Butantan Institute (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: NCV-02-IB
Record Dates: First submitted 2022-04-27; First posted 2022-04-29 (Actual); Last update posted 2025-02-06 (Actual); Status verified 2024-02

CONDITIONS: Coronavirus Infections; Healthy
Keywords: Vaccine; SARS-CoV-2; COVID-19
MeSH Terms: conditions — Coronavirus Infections; COVID-19 | interventions — NDV-HXP-S COVID-19 vaccine; BNT162 Vaccine

STUDY DESIGN:
Intervention Model Description: Parallel Assignment in Phase II (1:1), that aims to evaluate safety and immunogenicity in 400 subjects. Phase III (3:1), that aims to evaluate safety in total population (n=4.000, 3000 in arm of NDV-HXP-S 10μg, 1000 subjects per each consecutive batch, and 1000 subjects in the active control arm), immunogenicity in a subcohort (n=1000) and consistency of three consecutive batches in part of the subcohort of immunogenicity correspondent only to the NDV-HXP-S 10μg arms (n=750).
Who Masked: Participant, Care Provider, Investigator
Masking Description: An electronic central randomization system will be used to designate the investigational product (IP) that each participant must receive. A team study non-blind, qualified member (nurse/pharmacist) will obtain the corresponding randomization, will separate the respective IP, will blind the product and deliver it to blind staff. The product will be in a syringe that is in a blister labeled with the sponsor's name, IP code, administration route, IP dose and expiration date. The study non-blind staff will not have contact with the participants, will not have access to identification data or any other involvement with the study, besides randomizing the participant, separating the syringe containing active control or vaccine, checking if the information on the blister label corresponds the information on the cartridge label and the syringe is labeled with the clinical trial code, ID, corresponding visit and investigator's name.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (6):
- NDV-HXP-S 10μg (Phase II) (Experimental): In the Phase III, 200 adult subjects will be assigned to receive NDV-HXP-S 10μg/0.5mL intramuscular (deltoid), booster, 1 dose. All the population will be evaluated for safety and immunogenicity.
  Interventions: Biological: NDV-HXP-S 10μg
- BNT162b2 30μg (Phase II) (Active Comparator): In the Phase III, 200 adult subjects will be assigned to receive vaccine against COVID-19 BNT162b2 30μg/0.3mL intramuscular (deltoid), booster, 1 dose. All the population will be evaluated for safety and immunogenicity.
  Interventions: Biological: BNT162b2 30μg
- NDV-HXP-S 10μg batch 1 (Phase III) (Experimental): In the Phase III, 1000 adult subjects will be assigned to receive the first consecutive batch of NDV-HXP-S 10μg/0.5mL intramuscular (deltoid), booster, 1 dose. All the population will be evaluated for safety. Of them, 250 will be evaluated for immunogenicity and consistency of batches.
  Interventions: Biological: NDV-HXP-S 10μg
- NDV-HXP-S 10μg batch 2 (Phase III) (Experimental): In the Phase III, 1000 adult subjects will be assigned to receive the second consecutive batch of NDV-HXP-S 10μg/0.5mL intramuscular (deltoid), booster, 1 dose. All the population will be evaluated for safety. Of them, 250 will be evaluated for immunogenicity and consistency of batches.
  Interventions: Biological: NDV-HXP-S 10μg
- NDV-HXP-S 10μg batch 3 (Phase III) (Experimental): In the Phase III, 1000 adult subjects will be assigned to receive the third consecutive batch of NDV-HXP-S 10μg/0.5mL intramuscular (deltoid), booster, 1 dose. All the population will be evaluated for safety. Of them, 250 will be evaluated for immunogenicity and consistency of batches.
  Interventions: Biological: NDV-HXP-S 10μg
- BNT162b2 30μg (Phase III) (Active Comparator): In the Phase III, 1000 adult subjects will be assigned to receive the vaccine against COVID-19 BNT162b2 30μg/0.3mL intramuscular (deltoid), booster, 1 dose. All the population will be evaluated for safety. Of them, 250 will be evaluated for immunogenicity only.
  Interventions: Biological: BNT162b2 30μg

INTERVENTIONS:
Biological: NDV-HXP-S 10μg — NDV-HXP-S 10μg/0.5mL intramuscular (deltoid), 1 dose (booster)
  Arms: NDV-HXP-S 10μg (Phase II); NDV-HXP-S 10μg batch 1 (Phase III); NDV-HXP-S 10μg batch 2 (Phase III); NDV-HXP-S 10μg batch 3 (Phase III)
Biological: BNT162b2 30μg — Vaccine against COVID-19 BNT162b2 30μg/0.3mL intramuscular (deltoid), 1 dose (booster)
  Arms: BNT162b2 30μg (Phase II); BNT162b2 30μg (Phase III)

SUMMARY:
NDV-HXP-S is an inactivated COVID-19 vectored-vaccine virus using the Newcastle Disease Virus as basis and expressing Spike (S) protein from SARS-CoV-2 stabilized in pre-fusion form with Hexapro technology.

This vaccine was successfully tested in non-clinical and clinical studies with a good safety profile and eliciting neutralizing antibodies against SARS-CoV-2. Clinical testing is conducted by an international consortium including three different manufacturers. Butantan, in Brazil, is one of them.

DETAILED DESCRIPTION:
The present protocol of Phase II/III studies.The Phase II study consists in a randomized (1:1) controlled double-blinded trial that aims to evaluate the safety and immunogenicity of NDV-HXP-S 10μg as a dose of booster in comparison to the vaccine against COVID-19 BNT162b2 30μg in a population of 400 adult subjects (50% with age ≥ 60 years), regardless of past of infection by COVID-19, with proof of two or more doses of COVID-19, of which the last dose administered at least 120 days ago.

The Phase III study consists in a randomized (3:1) controlled double-blinded trial that aims to evaluate the safety, immunogenicity and consistency of three consecutive batches of NDV-HXP-S 10μg as a dose of booster in comparison to the vaccine against COVID-19 BNT162b2 30μg in a population of 4000 adult subjects (20% with age ≥ 60 years), with similar characteristics as the population of Phase II.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years, of which 50% and 20% were aged ≥60 years in Phase II and Phase III studies, respectively, regardless of previous SARS-CoV-2 infection status, with proof of four doses of any monovalent vaccine against COVID-19, of which the last dose administered at least 120 days to 540 days ago.
2. If pre-existing medical conditions: be in a stable condition that does not require hospitalization or significant changes in therapy during the three months prior to enrollment.
3. Agree to regular contact by phone, electronic means, and/or home visits.
4. Intention to participate in the study, documented by the Informed Consent Form.

Exclusion Criteria:

1. Administration of a vaccine of active or inactivated virus not provided for in the study regimen up to 30 days before the dose of the study vaccine.
2. Use of other COVID-19 vaccination regimen other than the one contemplated in item a. of the inclusion criteria.
3. Angioedema or anaphylactic reaction to previous immunizations.
4. Allergy to egg or chicken.
5. Severe allergic reaction or anaphylaxis to the vaccine or components of the study vaccine.
6. Suspected or confirmed fever within 24 hours prior to vaccination or an axillary temperature greater than 37.8°C* on the day of vaccination (inclusion may be delayed until the subject is fever-free for 24 hours), as well as confirmation of SARS-CoV-2 infection (enrollment should be deferred until the participant has completed 24 hours without fever or until the participant resolves the SARS-CoV-2 infection documented by two negative RT-PCR tests).
7. Evidence of uncontrolled active neurological, cardiac, pulmonary, liver or kidney disease. Significant treatment changes or hospitalizations for worsening the condition in the last three months are indicators of uncontrolled disease.
8. Bleeding disorders (e.g., clotting factor deficiency, coagulopathy, platelet dysfunction), or previous history of significant bleeding or bruising after intramuscular injection or venipuncture.
9. Neoplastic diseases (except basal cell carcinoma and cervical carcinoma in situ) diagnosed or under investigation.
10. Suspected or confirmed immune compromising diseases including congenital or acquired immunodeficiencies and autoimmune diseases not under control according to the medical history or physical examination, including asplenia. Significant treatment changes or hospitalizations for worsening the condition in the last three months are indicators of uncontrolled disease.
11. Use of immunosuppressive therapies six months prior to study inclusion or scheduled to be of service within two years of inclusion. The dose of corticosteroid considered immunosuppressive is the equivalent of prednisone at a dose of 20 mg/day for adults for more than 14 days. Continued use of topical or nasal corticosteroids and other topical immunomodulators or immunosuppressants will not be considered immunosuppressive. The following are considered immunosuppressive therapies: antineoplastic chemotherapy, radiotherapy, immunosuppressants to induce transplant tolerance, immunosuppressive and immunobiological treatments in patients with autoimmune rheumatic diseases, among others.
12. Use of blood products (transfusions or immunoglobulins) within the last three months prior to study inclusion or scheduled blood product or immunoglobulin administration within six months of study inclusion.
13. Alcohol or drug abuse in the past 12 months prior to the subject's inclusion.
14. Behavioral, cognitive, or psychiatric illness that affects the subject's ability to understand and cooperate with the study protocol requirements.
15. Being team member conducting the study or having a dependent relationship with one of the study team members.
16. Any other condition that may jeopardize the safety or rights of a potential participant or prevent him/her from complying with this protocol.
17. Abnormalities in screening laboratory tests are considered to be excludable in the opinion of the principal investigator or his/her medical representative. If any changes in the tests are considered temporary, the tests may be repeated up to three times during the screening period (Phase II only)
18. Positive serology tests for human immunodeficiency virus (anti-HIV1/2 ELISA); Hepatitis B (HbsAg or Anti-HBc) or Hepatitis C (total Anti-HCV ELISA).
19. Any other findings that the investigator expect to would increase the risk of adverse outcomes from study participation.

    For women of childbearing potential:
20. Pregnancy (confirmed by positive β-hCG test), being a breastfeeding, and/or manifest intention to have sexual practices with reproductive potential without the use of a contraceptive method (abstinence, sterilization, intrauterine or implantable contraceptive device; oral contraceptives; diaphragm or condom in combination with contraceptive gel, cream, or foam) within 30 days before and 28 days after vaccination.

    * Note: * The temperature measured with a temporal scanner skin thermometer is considered equivalent to the axillary temperature.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 4400 (Actual)
Dates: Start 2023-02-28 (Actual); Primary Completion 2023-10-05 (Actual); Study Completion 2024-09-25 (Actual)

PRIMARY OUTCOMES:
Solicited and unsolicited adverse reactions | Within to 7 days after vaccination booster dose
  Frequency and intensity of local and systemic solicited and unsolicited adverse reactions.
Unsolicited adverse reactions | Within 28 days after vaccination booster dose
  Frequency and intensity of all unsolicited grade ≥2 adverse reactions.
Severe adverse events | Within 28 days after vaccination booster dose
  Frequency, intensity and relatedness of severe adverse events.
Neutralization GMTR SARS-CoV-2 pseudovirus | Up to 28 days after vaccination booster dose
  Neutralization of Geometric mean titer ratio (GMTR) SARS-CoV-2 pseudovirus.
Seroconversion Neutralization GMT SARS-CoV-2 pseudovirus | Up to 28 days after vaccination booster dose
  Percentage of subjects with Seroconversion Neutralization GMT SARS-CoV-2 pseudovirus.

SECONDARY OUTCOMES:
GMT SARS-CoV-2 pseudovirus | Up to 28 days after vaccination booster dose
  Neutralization of Geometric mean titer (GMT) SARS-CoV-2 pseudovirus.
Neutralization GMFR SARS-CoV-2 pseudovirus | Up to 28 days after vaccination booster dose
  Neutralization Geometric mean fold rise ratio (GMFR) SARS-CoV-2 pseudovirus.
GMTR against SARS-CoV-2 (ELISA) | Up to 28 days after vaccination booster dose
  Geometric mean titer ratio (GMTR) of Anti-SARS-CoV-2-S IgG antibodies (ELISA).
Seroconversion anti-SARS-CoV-2 ELISA | Up to 28 days after vaccination booster dose
  Percentage of subjects with seroconversion of Anti-SARS-CoV-2 S IgG antibodies (ELISA).
GMFR against SARS-CoV-2 (ELISA) | Up to 28 days after vaccination booster dose
  Geometric mean fold rise ratio (GMFR) of Anti-SARS-CoV-2-S IgG titers (ELISA).
GMT against SARS-CoV-2 (ELISA) | Up to 28 days after vaccination booster dose
  Geometric mean titer (GMT) of Anti-SARS-CoV-2-S IgG antibodies (ELISA).
GMT against SARS-CoV-2 (ELISA) | Up to 3 and 12 months after vaccine booster dose
  Geometric mean titer (GMT) of Anti-SARS-CoV-2-S IgG antibodies (ELISA).
Neutralization GMT against SARS-CoV-2 pseudovirus (variants of concern) | Up to 28 days after vaccination booster dose
  Neutralization of Geometric mean titer (GMT) against SARS-CoV-2 pseudovirus (variants of concern)
T cell-mediated response against SARS-CoV-2 | Up to 12 months after vaccine booster dose
  Vaccine-induced T cell immune response against SARS-CoV-2 (parental and variants of concern) by AIM (Activation-Induced Marker) and electrochemiluminescence Meso Scale Discovery® (MSD) V-PLEX Human Biomarker.
Serious adverse events | Up to 12 months after vaccine booster dose
  Frequency, intensity and relatedness of serious adverse events.
Adverse events of special interest | Up to 12 months after vaccine booster dose
  Frequency, intensity and relatedness of adverse events of special interest.
Unsolicited adverse events | Up to12 months after vaccine booster dose
  Frequency and intensity of all unsolicited adverse events.
Hematologic and biochemical assessments (Phase II) | Up to 7 days after vaccine booster dose
  Frequency, severity and relatedness of hematologic (hemoglobin, white blood cells and platelets) and biochemical (AST, ALT, bilirubins and creatinine) out of reference values.
Adverse events with medical attention | Up to 12 months after vaccine booster dose
  Frequency, intensity and relatedness of adverse events with medical attention.

OTHER OUTCOMES:
Confirmed COVID-19 cases | From 14 days after booster to up to 12 months after vaccine booster dose
  Virologically confirmed COVID-19 cases 2 weeks after the booster
Possible case of VAERD | From 14 days after booster to up to 12 months after vaccine booster dose
  Possible cases of vaccine-associated enhanced respiratory disease (VAERD)

CONTACTS AND LOCATIONS:
Locations (6):
- Brazil (6):
  - Instituto Aggeu Magalhães - Fundação Osvaldo Cruz - Pernambuco, Recife, Pernambuco
  - Universidade Municipal de São Caetano do Sul, São Caetano do Sul, São Paulo
  - Centro de Pesquisa Clínica S, Serrana, São Paulo
  - Azidus Brasil Pesquisa Científica e Desenvolvimento Ltda., Valinhos, São Paulo
  - Instituto Lóbus, Volta Redonda, São Paulo
  - Instituto Brasil de Pesquisa Clínica (IBPClin), Rio de Janeiro

REFERENCES:
- [Derived] Nakahashi-Ouchida R, Fujihashi K, Kurashima Y, Yuki Y, Kiyono H. Nasal vaccines: solutions for respiratory infectious diseases. Trends Mol Med. 2023 Feb;29(2):124-140. doi: 10.1016/j.molmed.2022.10.009. Epub 2022 Nov 23. PMID 36435633